CLINICAL TRIAL: NCT01212614
Title: A Study for Measurement of Gastric Secretion by Magnetic Resonance Imaging (MRI) Under Inhibition of Gastric Secretion by Proton Pump Inhibitors in Healthy Subjects and Patients With Reflux Disease
Brief Title: Measurement of Gastric Secretion by MRI Under Inhibition by ProtonPump Inhibitors in Healthy Subjects & in GERD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KEK-ZH-Nr. 2010-0293
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Gastroesophageal Reflux Disease; Healthy Volunteers
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: MRI, non invasive 13C-breath test, 24h-intragastric / esophageal pH monitoring — MRI, non invasive 13C-breath test, 24h-intragastric/esophageal pH monitoring

SUMMARY:
This study bases on the successfully completed project SNF 320000-112006 (EK 1152 and SwissMedic 2005dr2207e) and will document the physiological effects of inhibited gastric secretion on the volume as well as the acidity of gastric secretion by high dose proton pump inhibitors in GERD patients and healthy controls. Twelve participants in each group will be studied in a randomized, double-blind placebo controlled trial. A novel non-invasive MRI technique developed in Zurich will assess the volume of gastric secretion following the ingestion of a regular liquid meal. In addition, intragastric / esophageal pH monitoring will assess the link between volume and intragastric distribution of gastric secretion on reflux events and symptoms. In addition, the effect of gastric secretion on outcome parameters of a non-invasive stable isotope breath test for measurement of gastric emptying will be assessed.

ELIGIBILITY:
Inclusion criteria: - Healthy volunteers must have less than one episode of reflux or dyspeptic symptoms per month of no more than mild severity in the last 3 months

- Reflux patients (GERD) must have chronic symptoms (>8 weeks) suggestive for GERD (definition and questionnaire see Appendix page 30). In addition, the initial screening manometry must show no severe esophageal dysmotility (e.g. spasm, achalasia). If in addition a pH-study has been performed the acid exposure must be > 4.2% / 24h.

Exclusion criteria: - Age under 18 or above 65

* Pathologic underweight or overweight (BMI < 18 or > 30 kg/m2)
* Previous history of gastrointestinal disease or surgery (excludes appendectomy, cholecystectomy, hernia repair and anorectal disorders)
* Previous cardiorespiratory (excludes arterial hypertension), hematologic, renal, atopic, alimentary or psychiatric disease, diabetes, drug or alcohol abuse
* Patient unable to stop medication that alters gut function for 72 hours prior to the study, including anticholinergics, prokinetics, proton-pump inhibitors, non-steroidal anti-inflammatory drugs
* Positive Helicobacter pylori status on 13C-Urea breath test
* Presence of metallic implants, devices or metallic foreign bodies
* Pregnancy and lactation (female patients of child bearing age will receive a pregnancy test prior to study)
* Female volunteers without adequate contraception for the duration of the study
* Involvement in any other clinical trial during the course of this trial, nor within a period of 30 days prior to its beginning or 30 days after its completion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To assess the volume of gastric secretion in GERD patients and healthy volunteers with and without acid suppression. | October 2010 - October 2012

CONTACTS AND LOCATIONS:
Overall Officials: Werner Schwizer, Professor MD, Principal Investigator — University Hospital Zurich, Gastroenterology and Hepatology
Locations (1):
- University of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Steingoetter A, Sauter M, Curcic J, Liu D, Menne D, Fried M, Fox M, Schwizer W. Volume, distribution and acidity of gastric secretion on and off proton pump inhibitor treatment: a randomized double-blind controlled study in patients with gastro-esophageal reflux disease (GERD) and healthy subjects. BMC Gastroenterol. 2015 Sep 2;15:111. doi: 10.1186/s12876-015-0343-x. PMID 26328588